CLINICAL TRIAL: NCT03923075
Title: The Effects of Dexmedetomidine on Induction of Anaesthesia and Onset of Neuromuscular Blockade in Children
Brief Title: Dexmetomidine in Children Undergoing General Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Paraskevi Matsota, Assoc Prof of Anaesthesiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DEXAINMBCH
Record Dates: First submitted 2019-04-16; First posted 2019-04-22 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2020-11

CONDITIONS: Anesthesia
Keywords: dexmedetomidine; propofol; rocuronium; TOF; children
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Drug: dexmedetomidine (Dexmed) solution(100μcg of dexmedetomidine in 50ml N/S 0.9%). given at a bolus dose of 0.5μcg/kg of the dexmedetomidine solution [that corresponds to the volume (ml) calculated by the type "body weight (Kg)/4 or body weight (Kg) X 0.25".
  THE SOLUTION IS GIVEN AS CONTINUOUS INFUSION 10 MINUTES BEFORE THE INDUCTION OF GENERAL ANAESTHESIA IN CHILDREN UNDERGOING ELECTIVE SURGERY
  Interventions: Drug: Dexmedetomidine
- 0.9 % saline (Placebo Comparator): Drug:0.9 % saline solution (Normal saline) given at a volume (ml) determined by the type: "body weight (Kg)/4 or body weight (Kg) X 0.25" THE SOLUTION IS GIVEN AS CONTINUOUS INFUSION 10 MINUTES BEFORE THE INDUCTION OF GENERAL ANAESTHESIA IN CHILDREN UNDERGOING ELECTIVE SURGERY
  Interventions: Other: 0.9% saline

INTERVENTIONS:
Drug: Dexmedetomidine — INFUSION BEFORE INDUCTION OF ANAESTHESIA
  Other Names: Dexmed
  Arms: Dexmedetomidine
Other: 0.9% saline — INFUSION BEFORE INDUCTION OF ANAESTHESIA
  Other Names: normal saline
  Arms: 0.9 % saline

SUMMARY:
The effects of dexmedetomidine on the onset of both the general anaesthesia induction and the neuromuscular blockade in children of school age will be investigated. Ten minutes before the induction of general anaesthesia, the first group will receive continuous infusion of dexmedetomidine (DEX group), while the second group will receive normal saline (Placebo group).

DETAILED DESCRIPTION:
Children 4 to 12 years old, ASA I-II, scheduled for elective minor or medium procedure under general anaesthesia will be included in the study, after written informed concern from their parents has been obtained. Participants will be randomly allocated according to the type of the solution infused 10 minutes before the induction of general anaesthesia into one of the following two groups using the closed envelop method.

DEX group: patients will receive 0.5μcg/kg IV bolus of dexmedetomidine in 10 min, right before the induction of general anaesthesia. The concentration of dexmedetomidine solution is 0.2μcg/ml, (100μcg of dexmedetomidine are diluted in 50ml N/S 0.9%), which corresponds to volume (ml) calculated by the type: "body weight (Kg)/4 or body weight (Kg) X 0.25".

Placebo group: patients will receive N/S 0.9% IV in 10 min, right before the induction of general anaesthesia. The volume infused (ml) is determined by the same type: "body weight (Kg)/4 or body weight (Kg) X 0.25".

The above solutions will be prepared by the anaesthetist who will provide the anaesthesia and will not be known to the anaesthetist who will record the study's measurements.

No premedication will be given. All children will receive the same anaesthesia induction scheme.

Once the patients have entered the operating theater, standard monitoring will be applied (NIBP, ECG, SpO2) and an IV line will be inserted. Depth of anaesthesia and monitoring of neuromuscular blockade will be recorded by BIS and TOF, respectively. Afterwards continues infusion of dexmedetomidine or N/S 0.9% will be initiated, depending on the assigned group, for duration of 10 min.

Right after the end of the infusion, we will proceed to the induction of anaesthesia with 3mg/kg of propofol and 2μcg/kg of fentanyl and when BIS<60 will be achieved, rocuronium will be administered at a dose of 0.7 mg/kg . Right afterwards, neuromuscular blockade will be estimated using the TOF acceleromyography (4 supramaximal twitches, 0.5sec interval in 2sec, frequency 2Hz, intensity 50mA). TOF will be repeated every 15sec. At the same time, ventilation of the patient will be supported with a bag and mask (Ο2 100%). When TOF=0 will be achieved, the patient will be intubated. After intubation, anaesthesia will be maintained with sevoflurane 1 MAC in 50% O2/Air.

The intubation conditions will be estimated using the Viby-Mogensen score (scale of 5 parameters). Also, number of intubation attempts will be recorded.

The study period is from "right before the start" of the dexmedetomidine or the N/S 0.9% infusion up to 5 min after the tracheal intubation. The following time points will be recorded:

Start time of the IV infusion of dexmedetomidine or N/S 0.9% (tstart) End time of the IV infusion of dexmedetomidine or N/S 0.9% (tend) Time of propofol injection (tprop) Time of achieving BIS<60 (tBIS<60) Time from propofol injection to achieve BIS<60 (tprop - tBIS<60) in min Time of rocuronium injection (troc) Time of achieving TOF=0 (tTOF=0) Time from rocuronium injection to TOF=0 (troc - tTOF=0) in min Time that intubation performed (tintubation)

Measurements Heart rate (HR), systolic arterial pressure (SAP), SpO2 and BIS will be recorded at the following time points: just before the start of infusion of dexmedetomidine or N/S 0.9% (tbaseline) and afterwards every 3 min during the infusion, as well as at the particular time points tend, tprop, tBIS<60, troc, tTOF=0, tintubation and 5 min after the intubation. Viby-Mogensen score and number of intubation attempts will also be recorded.

During the study period, any adverse effects or incidences like respiratory depression during the 10 min infusion of the study solutions, bradycardia (defined as >20% reduction of HR from the baseline values or as HR<60bpm), hypotension (defined as >20mmHg reduction of SAP from the baseline values), allergic reactions, bronchospasm and laryngospasm will be recorded. In case of bradycardia or hypotension, IV atropine 0.02μcg/kg or ephedrine 1-2μcg/kg will be administered, respectively. In case of persistent bradycardia despite the use of atropine, dexmedetomidine infusion will be stopped and the child will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* children underoing elective surgery under general anaesthsia
* age 4-12 years old
* ASA I-II

Exclusion Criteria:

* patient or parent refusal
* Mallampati score> 3
* BMI>35
* severe systemic cardiac disease
* neuromuscular disease
* recent respiratory infection
* drug allergy

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Onset of neuromuscular blockade | Up to 5 minutes after the injection of rocuronium
  Neuromuscular blockade is estimated with TOF acceleromyography, while onset of neuromuscular blockaded is defined as the time needed to achieve TOF=0 after the injection of rocuronium.

SECONDARY OUTCOMES:
Onset of anaesthesia induction | Up to 15 minutes after the initiation of the infusion of dexmedemoditine or normal saline, respectively
  The depth of anaesthesia is monitored using the BIS device (range 0-100). Onset of anesthesia is defined as the time needed to achieve BIS value<60, after the injection of propofol.
Number of participants who developed bradycardia | Up to 30 minutes after the initiation of the infusion of dexmedemoditine or normal saline, respectively
  Bradycardia is defined as >20% reduction of HR from the baseline values or as HR<60bpm using ECG monitoring.
Number of participants who developed hypotension | Up to 30 minutes after the initiation of the infusion of dexmedemoditine or normal saline, respectively
  Hypotension is defined as >20mmHg reduction of SAP from the baseline values using noninvasive monitoring of arterial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Georgia K Kostopanagiotou, Study Chair — 2nd Department of Anaesthesiology, "Attikon" University Hospital; Paraskevi K Matsota, Principal Investigator — 2nd Department of Anaesthesiology, "Attikon" University Hospital
Locations (1):
- 2nd Department of Anesthesiology, Attikon University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
restrictions due to regulation for personal data protection

REFERENCES:
- [Derived] Kouna N, Matsota P. Effect of Dexmedetomidine on Rocuronium-Induced Neuromuscular Blockade and Intubation Condition in Children: A Randomized Controlled Trial. Paediatr Anaesth. 2026 Mar;36(3):316-325. doi: 10.1002/pan.70098. Epub 2025 Dec 20. PMID 41420428